CLINICAL TRIAL: NCT00554047
Title: Effectiveness and Costs of Post-diagnosis Treatment in Dementia Coordinated by Multidisciplinary Memory Clinics in Comparison to Treatment Coordinated by General Practitioners
Brief Title: Comparison of Effectiveness and Costs of Post-diagnosis Treatment in Dementia
Acronym: AD-Euro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Netherlands Alzheimer Foundation (Other); Amsterdam UMC, location VUmc (Other); Maastricht University Medical Center (Other); Karolinska Institutet (Other); Stockholm Health Economics AB (Unknown); Slingeland Hospital (Other); Elkerliek Hospital (Other); Ggz Oost Brabant (Other); Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ADE 072510; ZonMw 80-007022-98-07703; ZonMw 945-07-7039
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-08

CONDITIONS: Dementia
Keywords: Dementia; Caregivers; Costs and cost analysis; Multicenter study; Randomized controlled trial; Quality Adjusted Life Years; Quality of life; Technology assessment, biomedical; Methods
MeSH Terms: conditions — Dementia | interventions — General Practitioners

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Multidisciplinary Memory Clinic
  Interventions: Other: Multidisciplinary Memory Clinic
- 2 (Active Comparator): General practitioner
  Interventions: Other: General Practitioners

INTERVENTIONS:
Other: Multidisciplinary Memory Clinic — Post-diagnosis treatment and coordination of care for patients with dementia and their informal caregivers delivered by Multidisciplinary Memory Clinics (MMCs)
  Arms: 1
Other: General Practitioners — Post-diagnosis treatment and coordination of care for patients with dementia and their informal caregivers delivered by general practitioners
  Arms: 2

SUMMARY:
In the Netherlands a rapidly increasing number of multidisciplinary memory clinics (MMC) currently diagnose 25% of the patients with dementia. Following the diagnostic work-up, MMCs are increasingly involved in post-diagnosis treatment and coordination of care, which probably is very important for patients and caregivers, but also very time consuming and expensive. This study will focus on the important question whether this complex post-diagnosis treatment and care coordination, evaluated both on effectiveness and costs, should be carried out by MMCs (intervention) or by General Practitioners (GPs) (control) as pivot of delivery of health care for these patients.

Objectives: To determine MMCs' effectiveness and cost-effectiveness in post-diagnosis treatment and care-coordination for dementia-patients and their caregivers compared to the post-diagnosis treatment and care coordination by GPs.

Time schedule: 12 months for including patients and their caregivers and 12 months of follow-up.

Annex Study: Specifically for the Health Technology Assessment (HTA) methodology study the main study will be extended with some experimental proxy measurements and alternative measurement approaches.

The objective of this Annex-study is to explore the feasibility and validity of Health Related Quality of Life (HRQL) value measurement in dementia patients. And to study the characteristics of proxy rating in HRQL research in dementia and the suitability and validity of yielding HRQL measurements by proxy assessment. Furthermore to explore the validity, reliability, and feasibility of the EQ5D and EQ6D in dementia research (in patients and in/by proxies); response shift, and alternative (more simple) methods of HRQL measurement and validate the Dutch versions of the QOL-AD and the use of the CarerQol-7D in dementia research.

ELIGIBILITY:
Inclusion Criteria:

* A patient with a new dementia diagnosis made at the MMC of the participating centre fulfilling DSM-IV-TR criteria with a CDR 0.5, 1 or 2
* Each patient has a caregiver
* Both patients and caregivers can provide informed consent for participation in the study

Exclusion Criteria:

* Life expectancy less than 1 year
* Living in a nursing home
* Already evaluated as being suitable for living in a nursing home
* Data collection impossible (e.g., due to severe visual/hearing/language impairment, mood disorder, or behavioral disturbances)
* The patient's general practitioner does not agree to participate
* Already participating in another study
* The patient visits the MMC for a second opinion
* Travel distance between MMC and patient's living address more than 50 kilometers
* A definite indication for memory clinic follow up:

  * A definite need for symptomatic drug treatment as judged by treating physician (e.g., Dementia with Lewy Bodies)
  * A definite need for specialist guidance as judged by treating physician (e.g., Creutzfeldt-Jakob Disease, severe Frontotemporal Lobar Disease)
  * A definite wish for symptomatic drug treatment by patient or caregiver
  * A definite need for guidance from psychiatric services involved in the memory clinic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-12; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Proxy-rated Health Related Quality of Life of the patient (cpQol-AD) | at 0, 6 and 12 months
Informal caregivers burden (Sense of competence (SCQ)) | at 0, 6 and 12 months
Cost utility analysis (EQ 5D) | at 0, 6 and 12 months

SECONDARY OUTCOMES:
Geriatric Depression Scale (GDS-15) | at 0, 6 and 12 months
Care-related quality of life of informal caregivers (CarerQol-7D + CarerQol-VAS) | at 0, 6 and 12 months
Quality of Live AD caregiver (cQoL-AD) | at 0, 6 and 12 months
Neuro Psychiatric Inventory (NPI-Q) | at 0, 6 and 12 months
Functional performance patient (IDDD) | at 0, 6 and 12 months
Patients rated Health Related Quality of Life (pQol-AD) | at 0, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. M. Olde Rikkert, MD PhD, Principal Investigator — University Medical Centre St Radboud, Nijmegen
Locations (9):
- Netherlands (9):
  - VU Medical Center, Alzheimer Centre, Amsterdam
  - Alysis Zorgroep, Rijnstate Hospital, Department of Geriatrics, Arnhem
  - GGZ Oost Brabant, Department of Geriatrics, Boxmeer
  - Slingeland Hospital, Department of Geriatrics, Doetinchem
  - Hospital Gelderse Vallei, Department of Geriatrics, Ede
  - Catharina hospital, Department of Geriatrics, Eindhoven
  - Elkerliek Hospital, Department of Geriatrics, Helmond
  - University Hospital Maastricht, Alzheimer Centre, Maastricht
  - University Medical Centre St Radboud, Alzheimer Centre, Nijmegen

REFERENCES:
- [Derived] Meeuwsen E, Melis R, van der Aa G, Goluke-Willemse G, de Leest B, van Raak F, Scholzel-Dorenbos C, Verheijen D, Verhey F, Visser M, Wolfs C, Adang E, Olde Rikkert M. Cost-effectiveness of one year dementia follow-up care by memory clinics or general practitioners: economic evaluation of a randomised controlled trial. PLoS One. 2013 Nov 25;8(11):e79797. doi: 10.1371/journal.pone.0079797. eCollection 2013. PMID 24282511
- [Derived] Meeuwsen EJ, Melis RJ, Van Der Aa GC, Goluke-Willemse GA, De Leest BJ, Van Raak FH, Scholzel-Dorenbos CJ, Verheijen DC, Verhey FR, Visser MC, Wolfs CA, Adang EM, Olde Rikkert MG. Effectiveness of dementia follow-up care by memory clinics or general practitioners: randomised controlled trial. BMJ. 2012 May 15;344:e3086. doi: 10.1136/bmj.e3086. PMID 22589500
- [Derived] Meeuwsen EJ, German P, Melis RJ, Adang EM, Goluke-Willemse GA, Krabbe PF, de Leest BJ, van Raak FH, Scholzel-Dorenbos CJ, Visser MC, Wolfs CA, Vliek S, Rikkert MG. Cost-effectiveness of post-diagnosis treatment in dementia coordinated by Multidisciplinary Memory Clinics in comparison to treatment coordinated by general practitioners: an example of a pragmatic trial. J Nutr Health Aging. 2009 Mar;13(3):242-8. doi: 10.1007/s12603-009-0066-1. PMID 19262961